CLINICAL TRIAL: NCT01870661
Title: Ultrasound Guided Peripheral Intravenous Catheter Insertion in the Hospitalized Patient: Long vs. Short Axis Placement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 035-13
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Need for IV Access
Keywords: Intravenous placement; Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long axis ultrasound placement of IV (Experimental): Long axis ultrasound placement of IV catheter
  Interventions: Device: Long axis IV placement with ultrasound
- Short axis ultrasound placement of IV (Active Comparator): Long axis ultrasound placement of IV catheter
  Interventions: Device: Short axis IV placement with ultrasound

INTERVENTIONS:
Device: Long axis IV placement with ultrasound — Peripheral IV placement with the ultrasound probe viewing the vessel in the long axis.
  Arms: Long axis ultrasound placement of IV
Device: Short axis IV placement with ultrasound — Peripheral IV placement with the ultrasound probe viewing the vessel in the short axis.
  Arms: Short axis ultrasound placement of IV

SUMMARY:
Comparison of peripheral IV catheters inserted by ultrasound using the long axis vs. the short axis technique. Our hypothesis is that long axis ultrasound placement will increase the longevity of the IV catheter.

ELIGIBILITY:
Inclusion Criteria:

* A patient who needs PIV access for intravenous medications and resuscitation either on a medical-surgical floor or in the ICU
* After floor team (including RN and/or house staff) and IV Nurse have attempted and failed or is not available

Exclusion Criteria:

* Need for vasopressors
* Need for TPN
* Need for hemodynamic monitoring
* Non English speaking patient
* Patients who are unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
catheter survival | 3 days
  How many catheters survived for 3 days or as long as they are needed.

SECONDARY OUTCOMES:
Need for central venous access | for 3 days
success rate of peripheral IV using ultrasound assistance | 30 minutes
Complication rate | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverberg, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Isreal Medical Center, New York, New York, United States